CLINICAL TRIAL: NCT06614998
Title: Establishment of an Early Warning Screening System for Hemophagocytic Lymphohistiocytosis: a Multi-center, Prospective Study
Brief Title: Establishment of an Early Warning Screening System for Hemophagocytic Lymphohistiocytosis a Multi-center, Prospective Study
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2024-KL100-01
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hemophagocytic Syndrome
Keywords: hemophagocytic syndrome screening system
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening patients with suspected hemophagocytic syndrome: Preliminary screening of patients with elevated ferritin and low fibrinogen, and then continue to improve triglycerides, abdominal color ultrasound and other examinations to further clarify, for some very suspicious patients, timely improve genes, NK cell activity and other tests, as soon as possible to determine whether they are patients with hemophagocytic syndrome
  Interventions: Drug: Patients diagnosed with HLH-94 should be treated as soon as possible

INTERVENTIONS:
Drug: Patients diagnosed with HLH-94 should be treated as soon as possible — For some highly suspicious patients, after diagnosis, according to the patient's etiology, the treatment plan should be determined as soon as possible, such as lymphoma-related patients treated with hormones combined with etoposide, which can greatly improve the prognosis of patients

SUMMARY:
Our three-step screening system uses commonly used clinical and laboratory parameters to effectively identify patients who may be at high risk of HLH, conduct etiology screening early for patients who meet the diagnostic criteria for HLH, and guide standardized treatment. Therefore, this study proposes to establish a highly accurate and convenient hemophagocytic early warning system to improve the early diagnosis of patients with hemophagocytic syndrome and identify suspected HLH patients early. Etiology screening is performed on patients who meet the diagnostic criteria for HLH, high-risk predisposing factors are identified, and precise treatment is guided, thereby improving the success rate of patient treatment and improving the quality of life.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Patients who meet the first step screening + have ≥ 3 abnormal screening indicators in the second step
2. Patients who meet the first step screening + have 2 abnormal screening indicators in the second step + patients with high-risk factors for HLH, such as history of lymphoma, EBV infection, autoimmune diseases, etc

Exclusion Criteria:

Exclusion Criteria Subjects who meet one of the following criteria will not be enrolled: 1. Patients with liver cirrhosis, liver cancer, and hepatic encephalopathy 2. Patients with trauma, hepatosplenic rupture and other organ hemorrhage 3. Patients with severe disease such as shock, sepsis, and multiple organ failure 4. Patients with DIC 5. Patients with long-term anemia 6. Patients with acute promyelocytic leukemia 7. Patients with idiopathic deafness 8. Patients who have taken hormones/immunosuppressants 72 hours before admission 9. Hereditary fibrinogen deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A three-step screening process identified 80 people with suspected hemophagocytic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The suspected patient was diagnosed with hemophagocytic syndrome after complete NK cell activity, triglyceride tests, etc. | Time forecasting:2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Affilitated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No